CLINICAL TRIAL: NCT03745716
Title: A Phase III Multicenter, Randomized, Open Label Study of APR-246 in Combination With Azacitidine Versus Azacitidine Alone for the Treatment of (Tumor Protein) TP53 Mutant Myelodysplastic Syndromes
Brief Title: APR-246 & Azacitidine for the Treatment of TP53 Mutant Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A18-15331
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: MDS
MeSH Terms: interventions — eprenetapopt; Azacitidine

STUDY DESIGN:
Intervention Model Description: This will be a Phase III, multicenter, randomized study to compare the rate of CR and duration of CR, in patients with TP53-mutated MDS who will receive APR-246 and azacitidine or azacitidine alone.
  Treatment will be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's disease.
  Patients will be randomized (1:1) to one of two arms: stratified by age (< 65 years versus ≥ 65):
  * Experimental arm: APR-246 + azacitidine; or
  * Control arm: Azacitidine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental arm: APR-246 + azacitidine (Experimental): Patients will be randomized (1:1) to one of two arms: stratified by age (< 65 years versus ≥ 65):
  Interventions: Drug: APR-246 + azacitidine
- Control arm: Azacitidine (Experimental): Patients will be randomized (1:1) to one of two arms: stratified by age (< 65 years versus ≥ 65):
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: APR-246 + azacitidine — Patients will be randomized (1:1) to one of two arms: stratified by age (< 65 years versus ≥ 65):
  Experimental arm: APR-246 + azacitidine; or Control arm: Azacitidine
  Arms: Experimental arm: APR-246 + azacitidine
Drug: Azacitidine — Patients will be randomized (1:1) to one of two arms: stratified by age (< 65 years versus ≥ 65):
  Experimental arm: APR-246 + azacitidine; or Control arm: Azacitidine
  Arms: Control arm: Azacitidine

SUMMARY:
A Phase III, multicenter, randomized study to compare the rate of complete response (CR) and duration of CR, in patients with TP53-mutated MDS who will receive APR-246 and azacitidine or azacitidine alone.

DETAILED DESCRIPTION:
A Phase III, multicenter, randomized study to compare the rate of CR and duration of CR, in patients with TP53-mutated MDS who will receive APR-246 and azacitidine or azacitidine alone.

Treatment will be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's disease.

Patients will be randomized (1:1) to one of two arms:

1. Experimental arm: APR-246 + azacitidine; or
2. Control arm: Azacitidine

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent (ICF) and is able to comply with protocol requirements
* Documented diagnosis of MDS, according to World Health Organization (WHO) classification
* Patient has adequate organ function as defined by the following laboratory values:

  1. Creatinine clearance > 30 mL/min (by Cockcroft-Gault method)
  2. Total serum bilirubin < 1.5 x Upper Limit of Normal (ULN) or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome or hemolysis or who required regular blood transfusions
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN
* Age ≥18 years at the time of signing the informed consent form (ICF)
* Having at least one TP53 mutation which is not benign or likely benign
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* If of childbearing potential, negative pre-treatment urine or serum pregnancy test
* If of childbearing potential (males and females), willing to use an effective form of contraception such as latex condom, hormonal birth control, intrauterine device or double barrier method during chemotherapy treatment and for at least six months thereafter

Exclusion Criteria:

* Patient has a known history of human immunodeficiency virus (HIV) or active hepatitis B or active hepatitis C infection (testing not mandatory)
* Patient has any of the following cardiac abnormalities (as determined by treating MD):

  1. Myocardial infarct within six months prior to registration,
  2. New York Heart Association Class II or worse heart failure (Appendix II) or known left ventricular ejection fraction (LVEF) < the institution lower limit of normal as assessed by echocardiogram
  3. A history of familial long QT syndrome,
  4. Clinically significant pericardial disease
  5. Electrocardiographic evidence of acute ischemia
  6. Symptomatic atrial or ventricular arrhythmias not controlled by medications
  7. QTc ≥ 470 msec (QT cardiac interval)
  8. Bradycardia (<40 bpm)
* Concomitant malignancies or previous malignancies with less than a 1-year disease free interval at the time of signing consent. Patients with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (e.g. cervix) may enroll irrespective of the time of diagnosis
* Prior exposure to azacitidine, decitabine or investigational hypomethylating agent
* Prior exposure to intensive chemotherapy
* Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of MDS within 14 days of the first day of study drug treatment
* No concurrent use of erythroid stimulating agents
* Patients with history of allogeneic stem cell transplantation
* Pregnant women are excluded from this study because APR-246 has not been studied in pregnant patients. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with APR 246, breastfeeding should be discontinued if the mother is treated with APR-246.
* Patients with active uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sallman, MD, PhD, Principal Investigator — Moffitt Cancer Center, Tampa, US
Locations (27):
- United States (23):
  - City of Hope, Duarte, California
  - Stanford University Cancer Research Center, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Health Care System South Florida, Hollywood, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Robert H Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University Of Chicago Medicine, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Holden Cancer Center, Iowa City, Iowa
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (4):
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Saint-Louis, Paris
  - IUCT Oncopole, Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: APR-246 + Azacitidine: APR-246 4.5mg/day (D1-4 of 28 day cycle) Azacitidine 75mg/m2 (D4-D10 of 28 day cycle)
- Control Arm: Azacitidine: Azacitidine 75mg/m2 (D4-D10 of 28 day cycle)
Period: Overall Study
Arm/Group | Experimental Arm: APR-246 + Azacitidine | Control Arm: Azacitidine
Started | 78 | 76
Completed | 75 | 74
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm: APR-246 + Azacitidine | Control Arm: Azacitidine | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 56 | 54 | 110
Age, Continuous [Median (Full Range); unit: years] | 69 [34 to 90] | 69.5 [29 to 86] | 69 [29 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 42 | 47 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 61 | 58 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  United States | 65 | 67 | 132
  France | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR)
Description: To compare the complete response rate, defined as the proportion of patients who achieve complete remission (CR) with APR 246 + azacitidine treatment vs. azacitidine only.
Time Frame: 12 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: APR-246 + Azacitidine | Control Arm: Azacitidine
Number analyzed (Participants) | 78 | 76
Participants | 27 | 17

ADVERSE EVENTS:
Time Frame: 12 months
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as adverse events that occurred after the first dose of study medication up to 30 days after last dose.
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 is used to grade severity of TEAEs. Severity Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life-Threatening, 5= Fatal.
  SAE and AE data reported for Safety Evaluable population. (Experimental Arm n=76; Control Arm n=61).
Arm/Group | Experimental Arm: APR-246 + Azacitidine | Control Arm: Azacitidine
All-Cause Mortality (participants affected / at risk) | 46/78 | 36/76
Serious Adverse Events (participants affected / at risk) | 53/76 | 38/61
Other Adverse Events (participants affected / at risk) | 76/76 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: APR-246 + Azacitidine (N=76) | Control Arm: Azacitidine (N=61)
Pneumonia (Infections and infestations) | 8 | 8
Sepsis (Infections and infestations) | 5 | 4
Septic shock (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Coronavirus infection (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Corynebacterium bacteremia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Escherichia bacteremia (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pseudomonal bacteremia (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sialadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal bacteremia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 14
Anemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 4
Asthenia (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Fecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hemorrhage intracranial (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 3
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Erythroleukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Vitreous hemorrhage (Eye disorders) | 1 | 0
Hemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: APR-246 + Azacitidine (N=76) | Control Arm: Azacitidine (N=61)
Constipation (Gastrointestinal disorders) | 48 | 32
Nausea (Gastrointestinal disorders) | 51 | 21
Vomiting (Gastrointestinal disorders) | 40 | 8
Diarrhea (Gastrointestinal disorders) | 23 | 17
Stomatitis (Gastrointestinal disorders) | 12 | 5
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Fatigue (General disorders) | 30 | 20
Pyrexia (General disorders) | 21 | 17
Injection site reaction (General disorders) | 16 | 17
Oedema peripheral (General disorders) | 18 | 14
Chills (General disorders) | 12 | 10
Anemia (Blood and lymphatic system disorders) | 33 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 16
Neutropenia (Blood and lymphatic system disorders) | 16 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 13
Neutrophil count decreased (Investigations) | 34 | 23
Platelet count decreased (Investigations) | 25 | 26
White blood cell count decreased (Investigations) | 31 | 29
Lymphocyte count decreased (Investigations) | 14 | 6
Headache (Nervous system disorders) | 24 | 13
Dizziness (Nervous system disorders) | 24 | 12
Paresthesia (Nervous system disorders) | 14 | 5
Tremor (Nervous system disorders) | 14 | 1
Hypokalemia (Metabolism and nutrition disorders) | 18 | 12
Decreased appetite (Metabolism and nutrition disorders) | 17 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 5
Hyponatremia (Metabolism and nutrition disorders) | 12 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 14 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Pneumonia (Infections and infestations) | 10 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Rash (Skin and subcutaneous tissue disorders) | 12 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 5
Insomnia (Psychiatric disorders) | 10 | 9
Confusional state (Psychiatric disorders) | 11 | 14
Anxiety (Psychiatric disorders) | 11 | 9
Hypotension (Vascular disorders) | 7 | 11
Hypertension (Vascular disorders) | 11 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 10
Fall (Injury, poisoning and procedural complications) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03745716/Prot_SAP_000.pdf